CLINICAL TRIAL: NCT04840381
Title: Dietary Habits and Lifestyle of Nonagenarians and Centenarians in the Italian Abruzzo Region
Status: Completed | Type: Observational
Sponsor: University of Teramo (Other)
Collaborators: DAngelino (Unknown)
Responsible Party: Principal Investigator, Mauro Serafini, Principal Investigator, University of Teramo
Other Study IDs: CenTEnari
Record Dates: First submitted 2021-03-10; First posted 2021-04-12 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: LONGEVITY 1; Diet Habit; Fasting; Activity, Motor
Keywords: Sdijuno; Centenarians; Dietary habits; Longevity; Fasting
MeSH Terms: conditions — Feeding Behavior; Fasting; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nonagenarians and Centenarians: Nonagenarians and Centenarians borned and living for most of their life in the Abruzzo region.
  Interventions: Behavioral: Questionnaire administrations

INTERVENTIONS:
Behavioral: Questionnaire administrations — Administration of an ad hoc questionnaire to register food frequency consumption and meal time, main recipes; phisical activity questionnaire and list of questions concerning the previous and actual health status of participants

SUMMARY:
The "CenTEnari" study is a cross-sectional study aiming at suveying the dietary and lifestyle habits of nonagenarians and centenarianss of citizens of the Abruzzo region, Italy.

DETAILED DESCRIPTION:
Several epidemiological studies indicates that diet and physical activity are two pivotal pillars for the maintenance the of the health status and for longevity. These two last factors seem to be strictly linked between them, as demonstrated by some studies on the so called "Blue zones", particular lands in the planet where longevity rate - in terms of nonagenarians and centenarians - is particularly high. In these studies, it has been pointed out that, other than genetics, individuals following dietary regimens with lower consumption of available carbohydrates and processed foods, higher consumption of fruit, vegetables, cereals and pulses and moderate intake of meat, fish and dairy foods live longer and in a healthier status.

The Abruzzo region is characterized by a great gastronomical variability, due also to the particular geographical characterization, with a few kilometer distance between sea and mountains. However, most of these dietary habits tend to stick in a valuable way to Mediterranean Diet, a dietary regimen listed in 2010 in the Representative List of the Intangible Cultural Heritage of Humanity by UNESCO. Intriguingly, the Mediterranean Diet is based on the intake of the above mentioned food groups, plus a recognized key role of the physical activity and conviviality in the meal consumption.

Particularly, in the internal and mountainous part of the Abruzzo region, it has been found that the local citizens followed/follows a typical "dietary practice" called "sdijuno", which in local dialect means "to break the fasting of the night". In fact, "sdijuno" was the first abundant meal of the day - usually at mid-morning, based on the local vegetable-based foods - following the previous frugal dinner and breakfast meals. Thus, it can be hypothesized of 14-16 hours of almost fasting period. This evidence falls into the most recent findings showing the importance to consume meals in the middle part of the day and limiting the caloric intake during evening time, when metabolism tends to decrease according to body circadian rhythm.

Based on these premises, the aim of the present study is to survey the dietary habits of nonagenarians and centenarians of the Abruzzo region - particularly focusing on their adherence to "sdijuno" practice - as well as physical activity and to collect personal data and health status information. Then, it will be investigated whether the adherence to the "sdijuno" dietary practice is relevant among the nonagenarians and centenarians and there is a link between this practice and the longevity of the volunteers. To do this, an ad hoc questionnaire has been set-up and will be administered to register food frequency and meal time, main recipes, physical activity habits, health status.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 90 years old
* Borned and living for most of their life in the Abruzzo region.

Exclusion Criteria:

* Age lower 80 years old.

Min Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Volunteers borned in the Abruzzo region and living in the Abruzzo region, or spent most of their life in the Abruzzo region.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Frequency of intake of food groups | 1 year
  Observed information regarding the frequency of the consumption different food groups during subejects' period of youth

SECONDARY OUTCOMES:
Moderate or Vigorous Physical Activity Per Week | 1 Week
  Self reported practice of moderate or vigorous physical activity per week during subejects' period of youth and old age (minutes-per-week)
Mealtime | 1 Day
  Self reported information regarding the daily mealtime during subejects' period of youth and old age (hour and minutes of meal eating)
Body weight | 1 Day
  Self reported body weight (kg)
Body height | 1 Day
  Self reported body height (m)
Body Mass Index (BMI) | 1 Day
  Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- University of Teramo - Faculty of Bioscience and Agro-Food and Environmental Technology, Teramo, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Angelino D, Godos J, Ghelfi F, Tieri M, Titta L, Lafranconi A, Marventano S, Alonzo E, Gambera A, Sciacca S, Buscemi S, Ray S, Galvano F, Del Rio D, Grosso G. Fruit and vegetable consumption and health outcomes: an umbrella review of observational studies. Int J Food Sci Nutr. 2019 Sep;70(6):652-667. doi: 10.1080/09637486.2019.1571021. Epub 2019 Feb 15. PMID 30764679
- [Background] Gensous N, Franceschi C, Santoro A, Milazzo M, Garagnani P, Bacalini MG. The Impact of Caloric Restriction on the Epigenetic Signatures of Aging. Int J Mol Sci. 2019 Apr 24;20(8):2022. doi: 10.3390/ijms20082022. PMID 31022953
- [Background] Magrone T, Perez de Heredia F, Jirillo E, Morabito G, Marcos A, Serafini M. Functional foods and nutraceuticals as therapeutic tools for the treatment of diet-related diseases. Can J Physiol Pharmacol. 2013 Jun;91(6):387-96. doi: 10.1139/cjpp-2012-0307. Epub 2013 Apr 12. PMID 23745830
- [Background] Poulain M, Pes GM, Grasland C, Carru C, Ferrucci L, Baggio G, Franceschi C, Deiana L. Identification of a geographic area characterized by extreme longevity in the Sardinia island: the AKEA study. Exp Gerontol. 2004 Sep;39(9):1423-9. doi: 10.1016/j.exger.2004.06.016. PMID 15489066